CLINICAL TRIAL: NCT03953612
Title: The Role of Neuroactive Steroids in Stress, Drug Craving and Drug Use in Cocaine Use Disorders
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1603017466; 1K01DA046561-01A1 (NIH)
Record Dates: First submitted 2019-04-24; First posted 2019-05-16 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Pregnenolone

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly assigned to 2 doses of PREG (300/500 mg/day) vs placebo (PLA) treatment (N=20/group) over 8 weeks.
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PREG 300 (Experimental): Eligible participants will be randomly assigned to PREG 300 mg/day over 8 weeks with a) an inpatient-outpatient option where they will be admitted to the Clinical Neuroscience Research Unit (CNRU) at the Connecticut Mental Health Center (CMHC) for first two weeks and then outpatient at Yale Stress Center (YSC) for the remaining 6 weeks, or b) an outpatient option where they will participate in the entire study outpatient at YSC.
  Interventions: Drug: Pregnenolone (PREG)
- patients receiving placebo (Placebo Comparator): Eligible participants will be randomly assigned to a placebo (PLA) treatment over 8 weeks with a) an inpatient-outpatient option where they will be admitted to the Clinical Neuroscience Research Unit (CNRU) at the Connecticut Mental Health Center (CMHC) for the first two weeks and then transition to outpatient at Yale Stress Center (YSC) for the remaining 6 weeks, or b) an outpatient only option where they will participate in the entire study outpatient at YSC.
  Interventions: Drug: Placebos
- PREG 500 (Experimental): Eligible participants will be randomly assigned to PREG 500 mg/day over 8 weeks with a) an inpatient-outpatient option where they will be admitted to the Clinical Neuroscience Research Unit (CNRU) at the Connecticut Mental Health Center (CMHC) for first two weeks and then outpatient at Yale Stress Center (YSC) for the remaining 6 weeks, or b) an outpatient option where they will participate in the entire study outpatient at YSC.
  Interventions: Drug: Pregnenolone (PREG)

INTERVENTIONS:
Drug: Pregnenolone (PREG) — 2 doses of PREG (300 or 500 mg/day)
  Arms: PREG 300; PREG 500
Drug: Placebos — placebo
  Arms: patients receiving placebo

SUMMARY:
To use pregnenolone (PREG; 300; 500mg) daily versus placebo (PLA) as a probe to assess the role of neuroactive steroids in individuals with cocaine use disorder (CUD).

DETAILED DESCRIPTION:
This experimental study aims to examine the effects of PREG on a) repeated cocaine craving, mood and neurobiological reactivity to brief, guided imagery exposure to stress, drug cues and neutral situations in the laboratory and b) daily cocaine intake, craving, cognition and mood in men and women with CUD; and c) sex differences in all of these outcomes. The study's hypothesis is that PREG vs PLA will dose-specifically decrease stress-induced and drug-cue induced cocaine craving, improve mood and cognitive performance, and normalize hypothalamic pituitary adrenal (HPA) axis response to stress and drug-cue imagery, and reduce cocaine intake and craving in daily life in individuals with CUD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals, ages 18 to 60.
* Subjects must meet current DSM-V criteria for cocaine use disorder; documented positive urine toxicology screen for cocaine at intake or collateral information from family members, significant others, room-mates etc., on recent use.
* Subject has voluntarily given informed consent and signed the informed consent document.
* Able to read English and complete study evaluations.

Exclusion Criteria:

* Women who are pregnant, or nursing or are of childbearing potential and not practicing an effective means of birth control.
* Meet current criteria for use disorder on another psychoactive substance, such as, heroin, amphetamines, hallucinogens/PCP, excluding alcohol and nicotine.
* Any current use of opiates or past history of opiate use disorder.
* Current use of any psychoactive drugs, including anxiolytics, antidepressants, naltrexone or antabuse.
* Any psychotic disorder or current Axis I psychiatric symptoms requiring specific attention, including need for psychiatric medications for current major depression and anxiety disorders.
* Significant underlying medical conditions such as cerebral, renal, thyroid or cardiac pathology which in the opinion of study physician would preclude patient from fully cooperating or be of potential harm during the course of the study.
* Abstinent from cocaine for more than two weeks prior to admission.
* Hypotensive individuals with sitting blood pressure below 90/50 mmHG.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Verica Milivojevic, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Stress Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PREG 300 mg/Day: Eligible participants will be randomly assigned to 300 mg/day PREG over 8 weeks with a) an inpatient-outpatient option where they will be admitted to the Clinical Neuroscience Research Unit (CNRU) at the Connecticut Mental Health Center (CMHC) for first two weeks and then outpatient at Yale Stress Center (YSC) for the remaining 6 weeks, or b) an outpatient option where they will participate in the entire study outpatient at YSC.
- PREG 500 mg/Day: Eligible participants will be randomly assigned to 500 mg/day PREG over 8 weeks with a) an inpatient-outpatient option where they will be admitted to the Clinical Neuroscience Research Unit (CNRU) at the Connecticut Mental Health Center (CMHC) for first two weeks and then outpatient at Yale Stress Center (YSC) for the remaining 6 weeks, or b) an outpatient option where they will participate in the entire study outpatient at YSC.
Period: Overall Study
Arm/Group | PREG 300 mg/Day | PREG 500 mg/Day | Patients Receiving Placebo
Started | 21 | 18 | 19
Intent to Treat Sample Included in Analyses | 20 | 17 | 18
Dropout Weeks 1-3 | 1 | 1 | 0
Dropout Weeks 4-12 | 1 | 0 | 0
Completed | 18 | 16 | 18
Not Completed | 3 | 2 | 1
Not completed — Randomized but did not start | 1 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PREG 300 mg/Day | PREG 500 mg/Day | Patients Receiving Placebo | Total
Number analyzed (Participants) | 20 | 17 | 18 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.05 (11.31) | 46.47 (11.06) | 47.17 (9.44) | 47.27 (10.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 6 | 16
  Male | 15 | 12 | 12 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 2 | 5
  Not Hispanic or Latino | 20 | 14 | 16 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 14 | 10 | 9 | 33
  White | 4 | 6 | 9 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 20 | 17 | 18 | 55
Years of Education [Mean (Standard Deviation); unit: years] | 12.5 (1.4) | 12.35 (1.87) | 12.56 (1.58) | 12.47 (1.59)
Number of Smokers [Count of Participants; unit: Participants] | 14 | 14 | 16 | 44

OUTCOME MEASURES:

1. Primary Outcome: Craving Change in Stress and Cue Relative to Neutral
Description: Cocaine craving assessed in a laboratory experiment with exposure to stress, cocaine cue and neutral control condition in those receiving PREG (300mg; 500mg) vs Placebo. Cocaine craving was assessed using the Cocaine Craving Questionnaire (CCQ), a brief 10-item self-report craving scale that ranges in mean score from 1 to 7, where a higher score indicates higher craving. Data presented here is craving change in stress relative to neutral and craving change in cue relative to neutral, where the possible range in mean change score is -6 to +6.
Time Frame: Experiment during treatment week 2
Population: A subset of participants from the full study sample completed the experimental component of stress and cocaine cue provocation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PREG 300 mg/Day | PREG 500 mg/Day | Patients Receiving Placebo
Number analyzed (Participants) | 8 | 11 | 11
score on a scale
  Stress Craving Change | 3.035 (1.34) | -0.486 (1.153) | 3.959 (1.115)
  Cue Craving Change | 0.031 (1.313) | -1.775 (1.126) | 4.835 (1.118)
Statistical Analysis 1: Comparison: PREG 300 mg/Day vs PREG 500 mg/Day vs Patients Receiving Placebo; Test type: Superiority; p < .001, Mixed Models Analysis; Linear mixed effects

2. Secondary Outcome: Anxiety Change in Stress and Cue Relative to Neutral
Description: Anxiety assessed in laboratory experiment with exposure to stress, cocaine cue and neutral control condition in participants receiving PREG (300mg; 500mg) vs. Placebo treatment. Anxiety was assessed using a 10-point visual analog scale (VAS) in which 0="not at all" and 10="extremely high", with the mean score ranging from 0 to 10, and where higher score means higher anxiety. Data presented here is anxiety change in stress relative to neutral and anxiety change in cue relative to neutral, where the possible range in mean change score is -10 to +10.
Time Frame: Experiment during treatment week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PREG 300 mg/Day | PREG 500 mg/Day | Patients Receiving Placebo
Number analyzed (Participants) | 8 | 11 | 11
score on a scale
  Stress Anxiety Change | 0.757 (0.309) | 0.118 (0.269) | 1.334 (0.263)
  Cue Anxiety Change | -0.305 (0.302) | 0.199 (0.261) | 0.959 (0.265)
Statistical Analysis 1: Comparison: PREG 300 mg/Day vs PREG 500 mg/Day vs Patients Receiving Placebo; Test type: Superiority; p < .001, Mixed Models Analysis; Linear mixed effects

3. Secondary Outcome: Cortisol Level Change in Stress and Cue Relative to Neutral
Description: Plasma was collected at each laboratory session to measure cortisol level and assess change in cortisol response to stress and cocaine cue relative neutral imagery condition exposure. Data presented here are change in cortisol level (mg/dl) in stress relative to neutral condition and cue relative to neutral condition.
Time Frame: Experiment during treatment week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | PREG 300 mg/Day | PREG 500 mg/Day | Patients Receiving Placebo
Number analyzed (Participants) | 8 | 11 | 11
mg/dl
  Stress Cortisol Level Change | -0.3 (0.55) | -0.52 (0.64) | 0.71 (0.9)
  Cue Cortisol Level Change | 0 (0.45) | -0.07 (0.73) | 0.58 (0.67)
Statistical Analysis 1: Comparison: PREG 300 mg/Day vs PREG 500 mg/Day vs Patients Receiving Placebo; Test type: Superiority; p = 0.7, Mixed Models Analysis; Linear mixed effects

4. Secondary Outcome: Pregnenolone Concentration
Description: Blood plasma concentration of pregnenolone in two doses of PREG (300mg; 500mg), and matching placebo, assessed over a 24 hour period.
Time Frame: between weeks 2-3 of treatment
Population: A subset of participants from the full study sample completed the experimental component of stress and alcohol cue provocation
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PREG 300 mg/Day | PREG 500 mg/Day | Patients Receiving Placebo
Number analyzed (Participants) | 8 | 11 | 11
ng/mL | 1.09 (0.194) | 1.54 (0.147) | 0.5 (0.146)
Statistical Analysis 1: Comparison: PREG 300 mg/Day vs PREG 500 mg/Day vs Patients Receiving Placebo; Test type: Superiority; p = 0.0001, ANOVA

5. Other Pre Specified Outcome: Cocaine Dollar Amount During Trial Period
Description: Mean dollar amount of cocaine per use day was assessed by daily self report on the Timeline Followback Substance Use Calendar and corroborated by daily self-reporting on smartphone (measurement unit in dollars).
Time Frame: up to 8 weeks
Population: Intent to Treat Sample Included in Analyses n=55
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | PREG 300 mg/Day | PREG 500 mg/Day | Patients Receiving Placebo
Number analyzed (Participants) | 20 | 17 | 18
dollars | 12.3 (17.57) | 26.44 (20.59) | 28.28 (43.99)
Statistical Analysis 1: Comparison: PREG 300 mg/Day vs PREG 500 mg/Day vs Patients Receiving Placebo; Test type: Superiority; p = 0.042, . Negative binomial regression models

6. Other Pre Specified Outcome: Mean Percent Cocaine Days
Description: The mean percent cocaine days as assessed by self report on daily smartphone monitoring and corroborated by the Timeline Followback Substance Use Calendar over the 8 week period.
Time Frame: up to 8 weeks
Population: Intent to Treat Sample Included in Analyses n=55
Measure: Mean (Standard Error); unit: percent days
Arm/Group | PREG 300 mg/Day | PREG 500 mg/Day | Patients Receiving Placebo
Number analyzed (Participants) | 20 | 17 | 18
percent days | 19.9 (20.46) | 35.12 (20.05) | 28.61 (26.19)
Statistical Analysis 1: Comparison: PREG 300 mg/Day vs PREG 500 mg/Day vs Patients Receiving Placebo; Test type: Superiority; p = 0.125, . Negative binomial regression models

ADVERSE EVENTS:
Time Frame: up to 8 weeks
Arm/Group | PREG 300 mg/Day | PREG 500 mg/Day | Patients Receiving Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 12/20 | 13/17 | 11/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PREG 300 mg/Day (N=20) | PREG 500 mg/Day (N=17) | Patients Receiving Placebo (N=18)
Dizziness (Nervous system disorders) | 1 | 0 | 0 — Lightheadedness
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PREG 300 mg/Day (N=20) | PREG 500 mg/Day (N=17) | Patients Receiving Placebo (N=18)
Headache (Nervous system disorders) | 2 | 2 | 3
Injury/Pain (General disorders) | 5 | 3 | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 1 | 1 — Gastrointestinal issues
Inflammation/Allergy (General disorders) | 1 | 1 | 1
Infection/Immune System (General disorders) | 2 | 3 | 1
Suicidal Thoughts (Psychiatric disorders) | 0 | 0 | 1
Lightheadedness (Nervous system disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 2 | 1 — Sleep Disturbance

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT03953612/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT03953612/ICF_001.pdf